CLINICAL TRIAL: NCT06295692
Title: A Phase 3, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of JNJ-77242113 for the Treatment of Participants With Generalized Pustular Psoriasis or Erythrodermic Psoriasis
Brief Title: A Study of JNJ-77242113 for the Treatment of Participants With Generalized Pustular Psoriasis or Erythrodermic Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 77242113PSO3005; 77242113PSO3005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Generalized Pustular Psoriasis; Erythrodermic Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-77242113- Participants With Generalized Pustular Psoriasis (GPP) or Erythrodermic Psoriasis (EP) (Experimental): Participants with GPP or EP will receive JNJ-77242113 tablet orally.
  Interventions: Drug: JNJ-77242113

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 tablet will be administered orally.

SUMMARY:
The purpose of this study is to evaluate how effective JNJ-77242113 is in participants with generalized pustular psoriasis (GPP) or erythrodermic psoriasis (EP).

ELIGIBILITY:
Inclusion Criteria:

* The study participant has a diagnosis of generalized pustular psoriasis (GPP) or erythrodermic psoriasis (EP) at screening. For GPP, a diagnosis must be classified based on the criteria for diagnosis of GPP by the Japanese Dermatological Association (JDA); for EP, has a history of plaque-type psoriasis. In addition, has an involved body surface area (BSA) of lesion greater than or equal to (>=) 80 percent (%) at baseline
* Candidate for phototherapy or systemic treatment for psoriasis (either naive or history of previous treatment)
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) at screening and have a negative urine pregnancy test at Week 0 prior to administration of study intervention
* A male participant must agree not to plan to father a child while enrolled in this study or within 90 days after the last dose of study intervention
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study intervention

Exclusion Criteria:

* The study participant has a total score of JDA severity index for GPP >=14 at baseline if participants have a diagnosis of GPP
* The study participant has a differential diagnosis of the erythroderma (for example, erythroderma caused by lymphoma or drug eruption) other than EP
* The study participant has a history of or current diagnosis or signs or symptoms of severe, progressive, or uncontrolled liver, renal; cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* The study participant has a history of amyloidosis
* Known allergies, hypersensitivity, or intolerance to JNJ-77242113 or its excipients
* The study participant who doesn't meet the criteria of prior/current concomitant therapy and/or history/conditions of infections

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2027-10-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (12):
- Japan (12):
  - JR Sapporo Hospital, Hokkaido
  - Ichinomiya Municipal Hospital, Ichinomiya
  - Teikyo University Hospital, Itabashi Ku
  - Hospital of the University of Occupational and Enviromental Health, Kitakyushu-shi
  - Kumamoto University Hospital, Kumamoto
  - Nagoya City University Hospital, Nagoya
  - Public Interest Incorporated Foundation Nipoon Life Saiseikai Nippon Life Hospital, Osaka
  - Tohoku University Hospital, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga Gun
  - Tokyo Medical University Hospital, Shinjuku
  - Fujita Health University Hospital, Toyoake
  - Mie University Hospital, Tsu

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are based on the primary completion date (14 Jan 2025). Remaining results will be reported within a year of study completion.
Groups:
- GPP: JNJ-77242113 200 mg QD: Participants with generalized pustular psoriasis (GPP) received JNJ-77242113 200 milligrams (mg) tablet orally once daily (QD) from Week 0 up to Week 24.
- EP: JNJ-77242113 200 mg QD: Participants with erythrodermic psoriasis (EP) received JNJ-77242113 200 mg tablet orally QD from Week 0 up to Week 24.
Period: Overall Study
Arm/Group | GPP: JNJ-77242113 200 mg QD | EP: JNJ-77242113 200 mg QD
Started | 9 | 10
Completed | 1 | 1
Not Completed | 8 | 9
Not completed — Ongoing | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GPP: JNJ-77242113 200 mg QD | EP: JNJ-77242113 200 mg QD | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (11.91) | 56.8 (14.01) | 58.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Generalized Pustular Psoriasis (GPP) Who Experienced Treatment Success at Week 16
Description: Percentage of participants with GPP who experienced treatment success at Week 16 was reported. Treatment success for GPP was defined as at least "minimally improved" rating in Clinical Global Impression (CGI) scale for GPP based on Japanese Dermatological Association (JDA) total score. JDA severity index includes skin symptoms (area of erythema with pustules, total area of erythema, and area of edema; each scored 0-3) and systemic/laboratory findings (fever, white blood cell count, C-reactive protein, and serum albumin; each scored 0-2). JDA total score was sum of 2 assessments ranging from 0 (best) to 17 (worst). CGI ratings were defined as: 1=Very much improved (greater than or equal to [>=]3-point reduction in JDA total score), 2=Much improved (1-2-point reduction), 3=Minimally improved (no change in JDA total score, but >=20 percent (%) reduction in area of erythema with pustules or meaningful improvement in >=1 other parameter), 4=No change, 5=Worsened. Higher score = worsening.
Time Frame: Week 16
Population: Full analysis set (FAS) included all enrolled participants who received at least 1 dose of JNJ-77242113. This outcome measure was planned to be analyzed for specified arm only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GPP: JNJ-77242113 200 mg QD
Number analyzed (Participants) | 9
Percentage of participants | 88.9 [51.8 to 99.7]

2. Primary Outcome: Percentage of Participants With Erythrodermic Psoriasis (EP) Who Experience Treatment Success at Week 16
Description: Percentage of participants with EP who experienced treatment success at Week 16 was reported. Treatment success for EP was defined as at least "minimally improved" rating in CGI scale for EP. The CGI scale is a clinician-rated 5-point scale with the following categories: 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Worsened. Higher score indicated worsening.
Time Frame: Week 16
Population: FAS included all enrolled participants who received at least 1 dose of JNJ-77242113. This outcome measure was planned to be analyzed for specified arm only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EP: JNJ-77242113 200 mg QD
Number analyzed (Participants) | 10
Percentage of participants | 100.0 [69.2 to 100.0]

3. Secondary Outcome: Percentage of Participants With GPP Who Experienced Treatment Success Over Time Based on CGI Scale According to JDA Total Score
Time Frame: From baseline (Week 0) to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

4. Secondary Outcome: Percentage of Participants With EP Who Experienced Treatment Success Over Time Based on CGI Scale
Time Frame: From Baseline (Week 0) to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

5. Secondary Outcome: Change From Baseline in the Total Score of the Japanese Dermatological Association (JDA) Severity Index for GPP Over Time
Time Frame: From baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

6. Secondary Outcome: Change From Baseline in Severity Classification of JDA Severity Index for GPP Over Time
Time Frame: From baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

7. Secondary Outcome: Change From Baseline in the Body Surface Area (BSA) of Involvement of Lesion for EP Over Time
Time Frame: From baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

8. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) Over Time
Time Frame: Baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

9. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of Cleared (0) Over Time
Time Frame: Baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

10. Secondary Outcome: Percent Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Over Time
Time Frame: From baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

11. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score Over Time
Time Frame: From baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

12. Secondary Outcome: Percentage of Participants Who Achieved DLQI Score of 0 or 1 Over Time
Time Frame: Baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

13. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension 5-Level (EQ-5D-5L) Over Time: Domain Scores
Time Frame: From baseline (week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

14. Secondary Outcome: Change From Baseline in EQ-5D-5L Over Time: Visual Analog Scale (VAS) Scores
Time Frame: From baseline (Week 0) up to Week 156
Reporting Status: Not Posted, anticipated posting 2028-10

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Time Frame: Baseline (Week 0) up to 160 weeks
Reporting Status: Not Posted, anticipated posting 2028-10

ADVERSE EVENTS:
Time Frame: From Week 0 up to Week 24
Description: Safety analysis set included all enrolled participants who received at least 1 dose of JNJ-77242113.
Arm/Group | GPP: JNJ-77242113 200 mg QD | EP: JNJ-77242113 200 mg QD
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/9 | 1/10
Other Adverse Events (participants affected / at risk) | 6/9 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GPP: JNJ-77242113 200 mg QD (N=9) | EP: JNJ-77242113 200 mg QD (N=10)
Acquired Haemophilia (Blood and lymphatic system disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GPP: JNJ-77242113 200 mg QD (N=9) | EP: JNJ-77242113 200 mg QD (N=10)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Keratitis (Eye disorders) | 1 | 0
Angular Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Oral Candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Suspected Covid-19 (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Carotid Arteriosclerosis (Nervous system disorders) | 0 | 1
Dizziness Postural (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Mechanical Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT06295692/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT06295692/SAP_001.pdf